CLINICAL TRIAL: NCT01862042
Title: Evaluation of Palliative and Supportive Care for Spinal Muscular Atrophy (SMA) Type 1 Patients
Brief Title: Palliative Care in Spinal Muscular Atrophy (SMA) 1
Acronym: ASI1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P110135; 2012-A00024-39 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2012-07-20; First posted 2013-05-24 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Spinal Muscular Atrophy 1
Keywords: Spinal Muscular Atrophy (SMA) type 1; Supportive care; Palliative care
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal | interventions — Surveys and Questionnaires; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive and Palliative care (Other): A follow-up diary will be completed by the families and the different practitioners working with the patient. One year after the death of the patient, a questionnaire will be proposed to the parents of the child by a psychologist.
  Interventions: Other: Follow-up diary and questionnaire

INTERVENTIONS:
Other: Follow-up diary and questionnaire — A follow-up diary will be completed by the families and the different practitioners working with the patient. One year after the death of the patient, a questionnaire will be proposed to the parents of the child by a psychologist.
  Other Names: Supportive and Palliative care

SUMMARY:
The purpose of this study is to evaluate the quality of supportive and palliative care for SMA type 1 patients.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy Type I (SMA I) is the most severe form of SMA. It presents in infancy and death occurs by 2 years. There is actually no curative treatment for this pathology. Support and help must be provided from the time of presentation till death and usually this period is quite short, about a couple of months. Variations in medical practice have be seen, depending on the medical experience and sometimes coupled with differences in family resources and values. The aim of the study is to evaluate the needs of the patients and their families, the medical practices, and to describe a cohort of SMA type 1 patients with the natural history of this disease. For this, a follow-up diary will be done, and this diary will be completed by the families and the different practitioners working with the patient. Will be noted in it : physical signs, all therapeutic choices and actions, evaluation of the pain and treatments. A special part of this follow-up diary will be completed by the medical doctors, after the death of the patient, with all the medication used at time of death and the conditions of the death. One year after the death of the patient, a questionnaire will be proposed to the parents of the child by a psychologist. This questionnaire will estimate the benefice of the follow-up diary, and the improvements to give in the diagnostic strategies, recommendations for assessment and monitoring, and therapeutic interventions in SMA type 1.

ELIGIBILITY:
Inclusion Criteria:

* SMA type 1 under 1 an
* Genetic confirmation

Exclusion Criteria:

* No genetic confirmation
* SMA type 1 over 1 year

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
%O2 | until 2 years
  Quantitative evaluation of care : oxygen therapy and Invasive ventilation

SECONDARY OUTCOMES:
Qualitative evaluation of the practices of care | until 2 years
  Analysis of the semi-structured questionnaire completed remotely by the methods of analysis semi-qualitative. Identification of the principal challenges faced by parents and satisfaction criteria or non-face to the proposed solutions.
Evaluation of nutritional status | until 2 years
  Quantitative evaluation of care : nutritional status and enteral nutrition
Evaluation of orthopedic facilities | until 2 years
  Quantitative evaluation of care : kinesitherapy and orthopedic facility
Evaluation of comfort | until 2 years
  quantitative evaluation of care : criterion for pain analgesics and sedatives care

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Desguerre, MD, PhD, Study Chair — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hully M, Barnerias C, Chabalier D, Le Guen S, Germa V, Deladriere E, Vanhulle C, Cuisset JM, Chabrol B, Cances C, Vuillerot C, Espil C, Mayer M, Nougues MC, Sabouraud P, Lefranc J, Laugel V, Rivier F, Louvier UW, Durigneux J, Napuri S, Sarret C, Renouil M, Masurel A, Viallard ML, Desguerre I. Palliative Care in SMA Type 1: A Prospective Multicenter French Study Based on Parents' Reports. Front Pediatr. 2020 Feb 18;8:4. doi: 10.3389/fped.2020.00004. eCollection 2020. PMID 32133329
- [Background] Ziegler HK, Unanue ER. Decrease in macrophage antigen catabolism caused by ammonia and chloroquine is associated with inhibition of antigen presentation to T cells. Proc Natl Acad Sci U S A. 1982 Jan;79(1):175-8. doi: 10.1073/pnas.79.1.175. PMID 6798568
- [Background] Kaufmann P, Greiss C, Brown J. Survival in SMA type 1. Neuromuscul Disord. 2009 Jan;19(1):76; author reply 76. doi: 10.1016/j.nmd.2008.10.010. Epub 2008 Dec 12. No abstract available. PMID 19070490
- [Background] Roper H, Quinlivan R; Workshop Participants. Implementation of "the consensus statement for the standard of care in spinal muscular atrophy" when applied to infants with severe type 1 SMA in the UK. Arch Dis Child. 2010 Oct;95(10):845-9. doi: 10.1136/adc.2009.166512. Epub 2009 Oct 8. PMID 19819869